CLINICAL TRIAL: NCT05983120
Title: The Effect of Education Provided According to Social Cognitive Learning Theory on Diabetes Self-management and Quality of Life in Individuals With Type 2 Diabetes Mellitus
Brief Title: Self-management and Quality of Life in Individuals With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yasemin Çelik, Dr. assistant professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Afyonkarahisar HSU
Record Dates: First submitted 2023-01-07; First posted 2023-08-09 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pre-Existing Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes; Social Cognitive Learning; Diabetes Self-management; Quality of Life
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): In the first five weeks, the experimental group was given training consisting of five modules, accompanied by power point presentations and applied social cognitive learning theory, then SMS reminders were sent every fortnight for seven weeks, and the study was completed at the end of the twelfth week. The control group received standard training from a diabetes nurse. Scale evaluations, metabolic and anthropometric measurements were made at the beginning and end of the study in the experimental and control groups. In addition, the scale evaluation was repeated in the fifth week for the experimental group. Data were evaluated using appropriate statistical methods.
  Interventions: Other: Education
- Control Group (No Intervention): The control group received standard training from a diabetes nurse.

INTERVENTIONS:
Other: Education — Educate the patients who suffer from Type 2 Diabetes Mellitus
  Arms: Training group

SUMMARY:
The study was conducted in order to study the effect of the training given according to social-cognitive learning theory (SCLT) upon diabetes self-management and quality of life among type 2 diabetes mellitus individuals.

DETAILED DESCRIPTION:
The study was done as a randomized-controlled experimental study at Internal Diseases Polyclinics of Afyonkarahisar Public Hospital between November 2021 and August 2022. The study was completed with 60 patients -experimental group (30 patients) and control group (30 patients)- who met inclusion criteria. The data were gathered using Information Request Form and Metabolic Variables Form, Diabetes Self-Management Scale (DSMS) for Type 2 Diabetic Patients, Multidimensional Scale of Perceived Social Support (MSPSS), Type 2 Diabetes Mellitus Self-Management Questionnaire (SMQ), WHOQOL-BREF (WHO- Quality of Life Scale- Short form). A theoretical and practical training based on SCLT was provided to the experimental group for the first five weeks -one module for each week- through power point presentations and afterwards, SMS reminders were sent every fifteen days for seven weeks and at the end of the twelfth week the training was completed. The control group received a standard training from diabetes nurse. The data were assessed using statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* Being diagnosed with Type 2 diabetes mellitus,
* Being on insulin therapy,
* Being open to verbal communication,
* Being literate
* Not to have an obstacle to continue the implementation phase of the research (for example, pregnancy plan, changing province, etc.)
* Not having hearing-vision problems and diabetes-related serious neuropathy (amputation, etc.),
* Patients who agreed to participate in the study.

Exclusion Criteria:The patient has a perception disorder and psychiatric disorder that prevents communication,

* Being pregnant,
* Individuals with serious complications such as retinopathy and neuropathy at the level of blindness were excluded from the study.

Research Termination Criteria

* Not performing the specified applications properly during the study,
* Unreachable in follow-ups,
* Those who want to quit working,
* Serious complications related to comorbid diseases and diabetes that occur during the working process,
* The study was terminated with patients who were moved out of the province during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Determination of self-regulation capacity from the principles of SCLT. | twelve weeks
  There is no specific score range.High scores on the scale indicate good self-management (SMQ), and low scores indicate poor self-management.
  In the intervention group, no significant change was observed in SMQ general score averages between PT2 and IT values compared to PT1. Similarly, no significant change was observed in PT2 values compared to PT1 regarding the control group score averages.
Determination of self-judgment capacity, one of the principles of SCLT. | twelve weeks
  DM was assessed with the Self-Efficacy Scale (DSMS). The lowest score that can be obtained from the scale is 20, and the highest score is 100. In the sample, the scale score average is calculated and individuals who are above the average are evaluated as high self-efficacy, and individuals below the average are evaluated as low self-efficacy.
  In the study, while the overall median score of DSMS in the intervention group showed a significant decrease in PT2 and IT values compared to PT1, no significant change was observed in the median DSMS scores of the control group.
Determining the effect of SCLT-based education on Quality of Life | twelve weeks
  Evaluated by WHOQOL - BREF (World Health Organization Quality of Life Scale - Short Form). It has four sub-dimensions: physical health such as pain, sleep, energy, psychological health such as positive emotions, self-confidence, body image, social relations such as social support, personal relations and environmental health such as economic status, transportation, safe environment and health conditions. A high score indicates a high quality of life.
  In the intervention group, no significant change was observed in the median values of physical health, psychological health, social relations, and environmental health, which are WHOQOL subscales, in PT2 and IT values compared to PT1. Compared to PT1 regarding the median score of the control group's social relations, a minimum significant increase was observed in PT2 values, but no significant change was found in other subscales

SECONDARY OUTCOMES:
Determination of blood HbA1c value. | twelve weeks
  HbA1c (glycosylated hemoglobin). Indicates the average blood glucose value over the last 2 to 3 months. The HbA1c reference range should be 5.7-6.4%. HbA1c level ≥6.5% or ≤5.6 poor glycemic control.
  In the intervention group, a significant decrease in the mean values of HbA1c, metabolic variables was observed compared to PT1 (9,53 ± 2,34) and PT2 ( 8,54 ± 1,77).
Determination of Fasting Blood Glucose (FBS) value. | twelve weeks
  It is the glucose value (plasma glucose) measured from a blood sample taken after eight or twelve hours of fasting. The normal reference range is min 80 mg/dl - max 130 mg/dl. FBS level ≥130 mg/dl or ≤80 mg/dl poor glycemic control.
  In the intervention group, a significant decrease in the mean values of FBS metabolic variables was observed compared to PT1 (224,77 ± 101,57) and PT2 (168,53 ± 65,27).
Determination of blood Postprandial Blood Glucose (PBS) value. | twelve weeks
  PBS is the plasma glucose value measured two hours after the start of food intake after an eight-hour fast. The reference range is 140-199 mg/dl. TKS ≥200 mg/dl or ≤139 mg/dl a weak glycemic control.
  Compared to PT1 (289,13 ± 114,06), the decrease in PBS mean values in PT2 (264,93 ± 91,55) were not significant change was found.
Determination of blood fasting lipid profile (total cholesterol, HDL-cholesterol, LDL-cholesterol, triglyceride) values. | twelve weeks
  A blood sample taken after eight or twelve hours of fasting is used to determine the fasting lipid profile (total cholesterol, HDL-cholesterol, LDL-cholesterol, triglyceride) values. Fasting lipid profile reference range is (Total cholesterol 20 - 200 mg/dl, High Density Lipoprotein (HDL) reference range is 35 - 65 mg/dl, Low Density Lipoprotein (LDL) reference range is 60 - 130 mg/dl, Triglyceride reference range is 20 - 203 mg/dl). Values less or higher than the specified values are considered as negative cholesterol levels.
  In the intervention group, a significant decrease in the mean values of total cholesterol was observed compared to PT1(192,87 ± 35,87) and PT2 (183,37 ± 36,26) measurements. Compared to PT1, although the decrease in LDL mean values and triglyceride median values in PT2 measurements were not significant, no significant change was found in the HDL value.

OTHER OUTCOMES:
Determining the principle of mutual determination from the principles of the social cognitive learning theory (SCLT) | twelve weeks
  It was evaluated with the Multidimensional Scale of Perceived Social Support (MSPSS). The lowest score that can be obtained from the entire scale is 12, and the highest score is 84. A high score indicates high perceived social support.
  In the intervention group, the social support (MSPSS) general score median values caused a significant and moderate increase in PT2 and İT values compared to PT1. No significant change was observed between the median scores of the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Celik, Principal Investigator — Afyonkarahisar Health Sciences University; Sibel Karaca Sivrikaya, Study Director — Balikesir University; Alper Emre Kurt, Study Chair — Afyonkarahisar goverment hospital; Sezen Yılmaz, Study Chair — Afyonkarahisar goverment hospital
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT05983120/Prot_000.pdf